CLINICAL TRIAL: NCT04316858
Title: A Prospective Randomized Trial in Comparison of Zero Calorie Carbonated Drink or Water as a Solvent in Sodium Phosphate for Colonoscopy
Brief Title: Randomized Trial Comparing Carbonated Drink With Water as a Solvent for Colonoscopy Solution
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Hina Noman, Senior Registrar, Surgical Unit III, Civil Hospital, Dow University of Health Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: HNoman
Record Dates: First submitted 2020-02-22; First posted 2020-03-20 (Actual); Last update posted 2020-03-20 (Actual); Status verified 2020-03

CONDITIONS: Colonoscopy
MeSH Terms: interventions — sodium phosphate; Water

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Water (Active Comparator): Water will be used as solvent for sodium phosphate
  Interventions: Drug: Sodium phosphate; Dietary Supplement: Water
- Zero calorie carbonated drink (Active Comparator): Zero calorie carbonated drink will be used as solvent for sodium phosphate
  Interventions: Drug: Sodium phosphate; Dietary Supplement: Zero calorie carbonated drink

INTERVENTIONS:
Drug: Sodium phosphate — 90ml of sodium phosphate will be added to 800ml of solvent( water or zero calorie carbonated drink) and taken in divided doses one day prior to procedure. Whole solution will be finished 3 -4 hours before colonoscopy.
  Other Names: Colonoscopy solution
Dietary Supplement: Water — 800 ml of water will be added to 90 ml of sodium phosphate to facilitate its intake by the patients preparatory to colonoscopy
  Arms: Water
Dietary Supplement: Zero calorie carbonated drink — 800 ml of zero calorie diet cola will be added to 90 ml of sodium phosphate to facilitate its intake by the patients preparatory to colonoscopy
  Other Names: Diet cola
  Arms: Zero calorie carbonated drink

SUMMARY:
This prospective randomized trial will be conducted in all patients undergoing elective colonoscopies from February 2020 to August 2020 in Dowites Operation Theater Endoscopy suite by surgical unit III, Civil Hospital Karachi. Patient will be select randomly based on inclusion criteria. Patients will be advised to take 90ml of sodium phosphate in 800ml solvent ( zero calorie soft drink and water). Patients will be nil per oral from midnight aside from clear liquids. Serum electrolytes, urea, creatinine will be measured after and before bowel preparation. Bowel preparation will be assessed by consultant during endoscopy. Questionnaire will be filled by PI for palatability, tolerance of solution, adverse effects, and willingness to repeat the preparation.

DETAILED DESCRIPTION:
This prospective randomized trial will be conducted in all patients undergoing elective colonoscopies from February 2020 to August 2020 in Dowites Operation Theater Endoscopy suite by surgical unit III, Civil Hospital Karachi. Patient will be select randomly based on inclusion criteria. Patients will be advised to take 90ml of sodium phosphate in 800ml solvent ( zero calorie soft drink and water). Patients will be nil per oral from midnight aside from clear liquids. Serum electrolytes, urea, creatinine will be measured after and before bowel preparation. Bowel preparation will be assessed by consultant during endoscopy. Questionnaire will be filled by PI for palatability, tolerance of solution, adverse effects, and willingness to repeat the preparation.

90ml of sodium phosphate will be added to 800ml of solvent and taken in divided doses one day prior to procedure. Whole solution will be finished 3 -4 hours before colonoscopy. The instructions about how to take the solution will be clearly explained at the time of booking. Complete Blood Count and hepatitis B and C screening as routine shall be done. All procedure will be carried out under monitored sedation by trained colorectal surgeon from the faculty

ELIGIBILITY:
Inclusion Criteria:

* • Age > 18 years

  * Non-emergency / non urgent colorectal diseases (IBD, suspected colonic polyps, colorectal cancer)
  * Screening Colonoscopy

Exclusion Criteria:

* Age <18 years Pregnancy Intestinal obstruction Unfit patient Acute or serious illness Coagulopathy Unwilling patients

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Palatability of the solution including willingness to repeat the preparation | This will be collected at the procedure appointment which is expected to be 2-3 hours in length. This time will be labelled as time 0 and will be noted once. T
  This will be assessed by a questionnaire to be filled by the patient on check-in for the colonoscopy procedure. It will be scored on a scale of 1 to 4 as excellent, good, satisfactory or bad; score 1 being excellent result.

SECONDARY OUTCOMES:
Degree of bowel cleanliness. | This will be collected at the procedure appointment which is expected to be 2-3 hours in length.
  This will be assessed by a questionnaire to be filled by the endoscopist after completion of endoscopy. It will assessed on a scale of 1 to 4 as excellent, satisfactory, poor or bad, with score 1 being the excellent.
Incidence of adverse effects. | This will be collected at the procedure appointment which is expected to be 2-3 hours in length. It will be noted once.
  This will be assessed by the reporting of adverse effects by the patients and laboratory evaluation of electrolytes prior to and after bowel preparation. These will be noted on a proforma and following side effects will be noted: Nausea/vomiting, bloating, cramps, or electrolyte abnormalities.
Completion time of preparation. | This will be assessed only once on check-in for the colonoscopy procedure.This will be collected at the procedure appointment which is expected to be 2-3 hours in length.
  This will be assessed in minutes on check-in for the colonoscopy procedure.

CONTACTS AND LOCATIONS:
Overall Officials: hina noman, fcps, Principal Investigator — dow university and health sciences
Locations (1):
- Dow University, Karachi, Sindh, Pakistan

REFERENCES:
- [Derived] Khan H, Memon AS, Abbasi MR, Samo KA, Agha JM, Rathore L, Saeed S. A prospective randomized trial to compare the effectiveness of zero calorie carbonated drink and water as a solvent in sodium phosphate for colonoscopy. J Pak Med Assoc. 2022 Mar;72(3):409-412. doi: 10.47391/JPMA.2344. PMID 35320215